CLINICAL TRIAL: NCT05001295
Title: STUDY ON THE EFFECTIVENESS OF AN ONLINE AEROBIC THERAPEUTIC EXERCISE PROGRAM FOR PATIENTS WITH LIMITATION OF PERSONALITY: RANDOMIZED CLINICAL TRIAL
Brief Title: ONLINE AEROBIC THERAPEUTIC EXERCISE PROGRAM FOR PATIENTS WITH LIMITATION OF PERSONALITY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1518010
Record Dates: First submitted 2021-08-05; First posted 2021-08-11 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2021-08

CONDITIONS: Borderline Personality Disorder
Keywords: Border personality disorder; Physiotherapy; Aerobic Exercise; Emotional Regulation; Teleassitence
MeSH Terms: conditions — Borderline Personality Disorder; Emotional Regulation | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Experimental)
  Interventions: Procedure: Physical Activity
- Daily Live (Placebo Comparator)
  Interventions: Procedure: Physical Activity

INTERVENTIONS:
Procedure: Physical Activity — Following the guidelines of NICE, the program to be followed by the IG is designed so that the intervention lasts 5 weeks, divided into 4 levels of progressive intensity, in which sessions of 30 to 45 minutes of aerobic exercise will be carried out 2 days a week. week.

SUMMARY:
Introduction: Borderline personality disorder is a serious mental illness with high prevalence and difficult to diagnose. BPD is characterized by unstable relationships, distorted sense of self, emotional instability and a strong impulsiveness with weak impulse control. Physiotherapy in mental health, currently being developed, is considered potentially effective in order to improve physical and mental health and the quality of life related to health.

Objective: The main objective of this study is to analyze the effect of an aerobic therapeutic exercise plan in the quality of life of patients with BDP.

Methodological design: A random controlled critical trial is going to be carried out. A sample of 50 participants diagnosed with BPD, aged 18 years and older, will be taken. They will be divided randomly in two groups: control group and treatment group. The treatment group will carry out a program of aerobic exercise twice a week for five weeks divided in four defined levels of variable length. The variables that will be compared before and after the intervention are: seriousness according to symptomatology, depression and anxiety level, emotion regulation difficulty, life quality level, physical condition level and ability of effort. After the intervention, the results will be analyzed by means of statistical processing based on the data obtained.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, diagnosed with Borderline Personality Disorder according to DSM-V with moderate-high severity who are admitted to a care center 24 hours a day.
* People over 18 years of age.
* People who do not perform scheduled physical exercise.
* Have electronic means (computer / tablet / mobile) with an internet connection, as well as the cognitive and motor skills necessary to carry out the proposed exercises.

Exclusion Criteria:

* People with intellectual or physical disabilities that prevent them from carrying out the intervention.
* People with heart or respiratory problems that prevent them from doing physical exercise.
* People who are legally incapacitated.
* Not meeting the inclusion criteria.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Border Line Symptom list BSL 23 | The evaluations will be carried out before and after the intervention to be able to compare the results after the completion of the marked exercise program.
  It is composed of 23 items that refer to the symptoms that the participant had the previous week, and must be answered using a 5-point Likert-type scale where 0 is never and 4 is a lot. The patient is considered to be in a mild state up to a score of 48, in a serious state between 49 and 62 and in a very serious state with a score greater than 63

SECONDARY OUTCOMES:
Quality of life SF-8 | The evaluations will be carried out before and after the intervention to be able to compare the results after the completion of the marked exercise program.
  he 8 items of the instrument cover the following scales: Physical function, Physical role, Body pain, General health, Vitality, Social function, Emotional role and Mental health. The items on the SF-8 are ordered in such a way that the higher the score, the better the health status. To calculate the score of the questionnaire, the items will have to be recoded so that they follow the gradient of "the higher the score, the better the health" and then calculate the sum of the items that make up the scale (raw score of the scale)
Beck Anxiety Inventory (BAI) | The evaluations will be carried out before and after the intervention to be able to compare the results after the completion of the marked exercise program.
  It consists of 21 items related to common anxiety symptoms. This inventory emphasizes the consequential physical aspects of anxiety during the past week and now. For correction, each item III.
  it is valued from 0 to 3 points according to the selected option (0 'not at all'-1' slightly'-2 'moderately'-3' severely '); To obtain the overall score, the total value of all the items will be added (in the event that any item has more than one option selected, the one with the highest score will be considered). The score range varies from 0 to 63. Minimal anxiety is considered to have a score between 0 and 7, mild anxiety between 8 and 15, moderate anxiety between 16 and 25 and severe anxiety a score equal to or greater than 26
Difficulty in emotional regulation (DERS) | The evaluations will be carried out before and after the intervention to be able to compare the results after the completion of the marked exercise program.
  consists of 28 items that are grouped into five subscales: emotional inattention (lack of emotional awareness), emotional rejection (non-acceptance of emotional experiences), everyday interference (difficulty in focusing on goal-centered behaviors when is emotionally activated) and emotional lack of control (difficulty controlling strong emotions). The minimum score for this scale is 23 and the maximum 135
The Beck Depression Inventory (BDI-II) | The evaluations will be carried out before and after the intervention to be able to compare the results after the completion of the marked exercise program.
  consists of 21 items with four alternative responses ordered from least to greatest severity. The instrument must be answered according to the state in which each participant has been in the last two weeks, including today. For its correction, each item is valued from 0 to 3 points according to the selected option (0-1-2-3); To obtain the global score, the total value of all the items will be added, obtaining a total score that can vary from 0 to 63.
Physical Function 30-Seconds Chair Stand Test | The evaluations will be carried out before and after the intervention to be able to compare the results after the completion of the marked exercise program.
  the strength, endurance, speed and mobility of the lower limbs, as well as the ability to response to change after a therapeutic exercise intervention. The transition from sitting to standing as a form of exercise can be used to determine the aerobic threshold in young, physically healthy individuals. The therapist in charge of the evaluation will count the number of times that the participant has stood up completely during the 30 seconds of the test

CONTACTS AND LOCATIONS:
Locations (1):
- Aurora Romero, Valencia, Spain